CLINICAL TRIAL: NCT05616650
Title: A Phase II Trial of Focal Ultrahypofractionated Stereotactic Radiation Therapy for the Treatment of Unifocal Prostate Cancer
Brief Title: Focal Therapy With Stereotactic Body Radiation Therapy (SBRT) for Patients With a Single Prostate Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000611; 000611-C
Record Dates: First submitted 2022-11-11; First posted 2022-11-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-07

CONDITIONS: Prostatic Neoplasms; Prostate Cancer; Prostate Adenocarcinoma
Keywords: Sbrt; PSMA; Targeted Pet Imaging; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Focal SBRT (Experimental): Focal SBRT to the tumor focus within the prostate, with response assessed by biopsy and imaging, including 18F-DCFPyL PET/CT.
  Interventions: Drug: 18F-DCFPyL; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: 18F-DCFPyL — Each participant will receive a single IV dose of 18F-DCFPyL by bolus injection. The target administered activity will be 6.5 mCi with a lower limit of 6 mCi; dose variations will be in accordance with the Nuclear Regulatory Commission (NRC) standard dose variation (i.e., 20%) permitted for diagnostic clinical studies.
Radiation: Stereotactic Body Radiation Therapy — Intensity modulated radiotherapy will be delivered to a dose of 26Gy in two fractions with the second fraction performed within 8 days of the first session.

SUMMARY:
Background:

The current standard treatment of prostate cancer is either surgery or radiation. Typically, this includes either the removal or radiation of the whole prostate gland. Many people now seek out focal therapy options to decrease the side effects of treatment. Until now, several forms of physical destruction with heat (thermal ablation), cold (cryotherapy), sound waves (HIFU), laser (FLA), and electrical energy (IRE). A new type of radiation (SBRT) may be an effective way to cure men of early-stage prostate cancer with fewer side effects than standard treatments.

Objective:

To see how people with untreated localized prostate cancer will respond to focal therapy with SBRT.

Eligibility:

People aged 18 years and older with untreated localized prostate cancer (prostate cancer which has not spread outside of the prostate gland).

Design:

* Participants will undergo screening including blood tests, an MRI, a PSMA PET/CT (18F-DCFPyL), and a biopsy.
* Small, non-radioactive, gold seeds about the size of a grain of rice will be placed in and/or around the tumor to help target the radiation treatment.
* Radiation (SBRT) will occur in 2 separate sessions about 1 week apart. No sedation is used, these sessions are painless. Each session will take about 1-2 hours. Participants can go home afterwards.
* Follow-up will continue for 2 years with repeat scans (MRI and PSMA PET/CT) and blood (PSA) tests.
* After two years, a biopsy will be done to understand the impact of this new treatment on prostate cancer.

DETAILED DESCRIPTION:
Background:

* Prostate cancer is the most common cancer among American men.
* The best current validated treatment options include whole gland radiotherapy and radical prostatectomy.
* Based on recent advances in imaging, focal ablative therapies are under investigation in attempts to deliver comparable rates of tumor control with less side effects.
* Thus far, focal therapies such as cryotherapy, high-intensity focused ultrasound, or focal laser ablation have resulted in poor local control with the exception of implanted radiation sources which have shown in-field control rates > 90%.
* As such, the proposed trial is designed to investigate the efficacy of a novel form of focal stereotactic body radiation therapy (SBRT) for the treatment of localized, unifocal prostate cancer.
* Prostate specific membrane antigen (PSMA) targeted PET imaging was recently FDA approved for imaging men with suspected prostate cancer metastases who are potentially curable by radiation or surgery. 18F-DCFPyL, a second generation PSMA PET agent that binds with high affinity to PSMA yet clears rapidly from the blood pool will be used in this study.

Objective:

-To determine whether localized, tumor-directed SBRT can produce biopsy-confirmed tumor response at 24 months in participants with unifocal prostatic adenocarcinoma.

Eligibility:

* Histologically confirmed, low or intermediate risk prostatic adenocarcinoma verified by biopsy.
* Unifocal prostate cancer defined as a single focus of prostate cancer on imaging which is correlated with a positive targeted biopsy.
* Age >= 18.
* No concurrent systemic Androgen Deprivation Therapy (ADT) is planned.

Design:

* This is a single-arm phase II trial designed to measure the efficacy of a novel application of SBRT guided with advanced prostate-specific imaging techniques.
* Participants will initially undergo a treatment planning CT, multiparametric MRI (mpMRI), 18F-DCFPyL PET/CT imaging, a biopsy, quality of life (QoL) questionnaires and laboratory evaluations. SBRT will be administered at 26Gy in two fractions on two separate days.
* Following completion of treatment, participants will be followed for up to 2 years through clinical evaluation, laboratory evaluations (including a complete blood count (CBC), prostate specific antigen (PSA) and testosterone measurements), QoL assessments, mpMRI, 18FDCFPyL PET/CT imaging, and a biopsy.
* The accrual ceiling is set to 42 participants with the goal of recruiting 30 evaluable participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically confirmed, low or intermediate risk prostatic adenocarcinoma verified by biopsy (NIH Laboratory of Pathology confirmation is required).
* Unifocal prostate cancer defined as a single focus of prostate cancer on MRI and PSMA PET/CT imaging which is correlated with a positive targeted biopsy.
* Age >=18 years.
* ECOG performance status <=2 (Karnofsky >60%).
* Men must agree to use highly effective contraception with their partner (barrier method of birth control; abstinence) for the duration of study participation and up to 120 days after the last radiation treatment.
* Ability of individual to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with NCCN high-risk prostate cancer features (Gleason score >=8, >cT2c, or PSA >= 20 ng/mL).
* Participants with prostate biopsies which show >= grade group 2 adenocarcinoma determined to be outside of the radiographically visible lesion (systematic biopsies which map to a radiographically detected lesion are not an exclusion criterion).
* Participants in whom concurrent systemic Androgen Deprivation Therapy (ADT) or chemotherapy is planned.
* Participants who are receiving any other investigational agents.
* Participants found to have pelvic or distant metastases on pre-treatment staging studies.
* Participants with an AUA-SI/IPSS score > 18.
* Participants who have previously received curative treatment for a prior or the current diagnosis of prostate cancer.
* Active urinary tract infection assessed by urinalysis.
* Human immunodeficiency virus (HIV)-infected individuals who are not on effective anti-retroviral therapy. Participants on anti-retroviral therapy with undetectable viral load within the 6 months prior to registration are eligible for this trial.
* Participants with hepatitis B virus (HBV) infection who have not been treated and cured.
* Participants with chronic HBV at screening must have an undetectable HBV viral load on suppressive therapy.
* Participants with hepatitis C virus (HCV) infection who have not been treated and cured.
* Participants with HCV infection who are currently on treatment, are eligible if they have an undetectable HCV viral load at screening.
* Anatomic relationship between the tumor and adjacent normal tissues judged to be unfeasible for the planned treatment by the PI.
* Participants with connective tissue diseases.
* Participants with radiation hypersensitivity syndromes.
* Ongoing active inflammatory bowel disease within the radiation field.
* Participants with prior medical comorbidity or surgical history involving the low pelvis which is expected to confer a high risk of toxicity to the experimental radiation regimen.
* Ineligibility or unwillingness to undergo a contrast-enhanced MRI due to inadequate renal function (eGFR < 30), severe claustrophobia, a weight above tolerance of the scanner (> 350 lbs.), a body size unable to fit into the scanner, or implanted devices incompatible with an MRI (implanted cardiac devices, surgical hardware, retained shrapnel, cerebral aneurysm clips, or other incompatible objects.
* Unwillingness to undergo an 18F-DCFPyL PET/CT or known allergy to the 18F-DCFPyL tracer.
* Contraindication or inability to undergo fiducial marker implantation.
* History of prior radiotherapy overlapping with the intended radiation field.
* Uncontrolled intercurrent illness, factors, or social situations that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | 2 years
  The primary objective of this trial is to determine the pathologic complete response rate on biopsy at two years in patients undergoing focal SBRT for prostate cancer. This will be defined by a negative biopsy at 2 years post-treatment.

SECONDARY OUTCOMES:
Longitudinal quality of life (QoL) | baseline and 1, 3, 6, 9, 12, 15, 18, 21, and 24 months after focal SBRT
  The QoL scores will be summarized at baseline and for each visit. Linear mixed effects model will be used to model quality of life scores at baseline, during and after treatment. Changes of QoL scores from baseline at each timepoint treatment will be calculated from the estimated linear mixed effect model.
PSA kinetics | 1 week and 1, 3, 6, 9, 12, 15, 18, 21, 24 months after focal SBRT
  The PSA kinetics scores will be summarized at baseline and for each visit. Linear mixed effects model will be used to model PSA kinetics at baseline, during and after treatment. Changes of PSA kinetics during and after treatment will be calculated from the estimated linear mixed effect model. In the rare case where PSA test is done on outside laboratory assay, a sensitivity analysis will be conducted to analyze PSA kinetics with and without outside values to determine whether outside laboratory measurement influenced results.
Nadir PSA | 1 week and 1, 3, 6, 9, 12, 15, 18, 21, 24 months after focal SBRT
  The nadir PSA (time to nadir PSA and value of nadir PSA) will be described for this cohort (median, mean, standard deviation, and range).
Absolute and relative fraction of free PSA to bound PSA | 1 week and 1, 3, 6, 9, 12, 15, 18, 21, 24 months after focal SBRT
  Descriptive statistics for the absolute amount and relative fraction of free PSA and bound PSA at the various timepoints detailed in 10.1 will be reported will be compared with baseline by paired Wilcoxon test.
Toxicity profile | During the focal SBRT period and 1, 3, 6, 9, 12, 18, 24 months after focal SBRT
  Descriptive statistics will be used to summarize the toxicity profile of focal SBRT of prostate cancer.
Rate of biochemical failure | 24 months after focal SBRT
  The rate of biochemical failure as defined by nadir PSA + 2.0 ng/mL at 24 months will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Krishnan R Patel, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers 2 years after the completion of the primary endpoint.@@@@@@If dbGaP is applicable: Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000611-C.html